CLINICAL TRIAL: NCT06047808
Title: A Feasibility Study Evaluating Storytelling Through Music Intervention with Bereaved Parents of Children with Cancer
Brief Title: Feasibility Study of the Storytelling Through Music Intervention with Bereaved Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Carolyn Phillips, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004111
Record Dates: First submitted 2023-06-06; First posted 2023-09-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Cancer; Grief; Well-Being, Psychological; Coping Strategies; Bereavement
MeSH Terms: conditions — Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Storytelling Through Music (Experimental): Participants will be randomized to either the "Storytelling Through Music" (STM) experimental arm or the waitlist control arm. STM is a six-week intervention that utilizes storytelling, reflective writing, self-care skills (i.e., breathing exercises, meditation, self-compassion, body scans), and songwriting. The intervention is delivered online and in a group setting. Online delivery provides convenience to participants, and the group setting provides an environment of people with shared experiences, which has been shown to decrease social isolation and feelings of being alone in their emotional experience. By the end of the intervention, participants will have written a short story and a song based on their story.
  Interventions: Behavioral: Storytelling Through Music
- Waitlist Control (No Intervention): Participants will receive the same "Storytelling Through Music" intervention once data collection from the experimental arm is complete.

INTERVENTIONS:
Behavioral: Storytelling Through Music — "Storytelling Through Music" is a six-week expressive arts intervention.
  Arms: Storytelling Through Music

SUMMARY:
The death of a child, at any age, is considered one of the most stressful life events a person can experience. In 2020, 11,050 children (under 15 years), 5,000 adolescents (15-19 years) and 60,000 young adults (20-39 years) were estimated to be diagnosed with cancer in the US. While the five-year survival is better for children than adults, over 10,000 children, adolescents, and young adults die from cancer in the US each year.1 Bereaved parents often experience intense and lasting psychological distress resulting in significantly higher morbidity and mortality compared to non-bereaved parents. Twenty-five percent of bereaved parents report new diagnoses of illnesses including prediabetes, anxiety and sleep disorders. Bereaved parents also experience psychological distress such as anxiety, post-traumatic stress disorder, and grief-related depressive symptoms that continue to be significant for years after a child's death. A recent study showed that nearly 33% of bereaved parents suffered from prolonged grief five years after their loss.6 Physiologically, studies show increased cortisol, immune, endocrine, and cardio biomarkers in people with prolonged grief. The death of a child can also affect family and social relationships resulting in decreased communication, feelings of isolation, absence of close social relationships and increased marital strain and divorce.

The purpose of this randomized controlled pilot study is to evaluate the feasibility of implementing a six-week multi-dimensional intervention, Storytelling Through Music (STM), with parents of children who have died from cancer. STM combines multiple modalities of expression (storytelling, writing, and music) to facilitate loss- and restoration-oriented coping by creating a legacy piece (self-written story paired with song) to facilitate continuing bonds with the deceased and find meaning.

DETAILED DESCRIPTION:
The death of a child, at any age, is considered one of the most stressful life events a person can experience. In 2020, 11,050 children (under 15 years), 5,000 adolescents (15-19 years), and 60,000 young adults (20-39 years) were estimated to be diagnosed with cancer in the US. While the five-year survival is better for children than adults, over 10,000 children, adolescents, and young adults die from cancer in the US each year. Bereaved parents often experience intense and lasting psychological distress resulting in significantly higher morbidity and mortality than non-bereaved parents. Twenty-five percent of bereaved parents report new diagnoses of illnesses, including prediabetes, anxiety, and sleep disorders. Bereaved parents also experience psychological distress, such as anxiety, post-traumatic stress disorder, and grief-related depressive symptoms that continue to be significant for years after a child's death. A recent study showed that nearly 33% of bereaved parents suffered from prolonged grief five years after their loss. Physiologically, studies show increased cortisol, immune, endocrine, and cardio biomarkers in people with prolonged grief. The death of a child can also affect family and social relationships resulting in decreased communication, feelings of isolation, absence of close social relationships, and increased marital strain and divorce.

The World Health Organization and the National Coalition for Hospice and Palliative Care (NCHPC) advocate that palliative care should not only improve the quality of life of patients but also extend into bereavement for families. The NCHPC bereavement guideline (7.5.1.c) states that bereavement interventions should include rituals that acknowledge loss and transition, provide opportunities for remembrance, and establish a sense of community. Researchers have examined the use of life review, dignity therapy, and remembrance with pediatric and adolescent patients, as well as bereaved family caregivers of spouses. However, to our knowledge, none have been conducted with bereaved parents. Despite the high risk of negative outcomes and national guidelines recommending bereavement care, the resources for bereaved parents are scarce. In a recent systematic review of intervention studies for bereaved parents, only fifteen interventions were identified. Of those studies, most lacked empirical evidence of effectiveness or alignment with key theoretical concepts. To increase the number of effective resources for this vulnerable and underserved population, interventions need to be developed and tested in order to promote health and disease prevention in this high-risk population.

Mechanisms of Coping with Parental Grief

Parental bereavement is complex because many personal, relational, and end-of-life circumstances affect bereavement, and individuals cope differently. Several factors are associated with prolonged grief and poorer psychosocial outcomes, including intra-personal (i.e., attachment style, sex, religious beliefs, age, history of mental health problems), inter-personal (i.e., social support, family, culture, religious practice, resources), and the unexpectedness of the loss. However, none of these factors are easily changed by interventions. Focusing on modifiable processes that mediate or moderate the adaptation trajectory in bereavement may be more beneficial. In bereaved adults, processes that mediate the relationship between risk factors and mental health outcomes include rumination, deliberate grief avoidance, emotional expression, cognitive appraisals, and meaning-making.

Meta-Affective and Meta-Cognitive Effects of Grief

A growing body of research suggests that self-compassion is positively associated with well-being and negatively associated with depression, anxiety, and post-traumatic stress. Self-compassion recognizes suffering as a universally shared human experience and teaches people to face their suffering non-judgmentally with a kind and mindful approach. Only one study has examined the influence of self-compassion on grief processing, showing a significant relationship between low self-compassion and the severity of complicated grief. Self-compassion may be beneficial in coping with grief because it is associated with engagement in, rather than avoidance of, painful thoughts, memories, and feelings. Furthermore, research on meta-cognition has shown that maladaptive coping strategies such as rumination are driven by metacognitive appraisals of an internal or external event. Meta-cognitive beliefs may keep bereaved people focused on loss issues, preventing them from integrating the loss into their lives and planning for the future.

Affective and Cognitive Effects of Expressive Arts

Expressive arts have been used to improve psychosocial well-being in people with cancer, adolescents with grief, veterans with post-traumatic stress disorder, and to aid bereavement among family caregivers. Yet, many of these studies lack methodological rigor. Interventions aimed at meaning-making are good for individuals at high risk for prolonged grief. Music has been used across cultures, and there is growing evidence that music is often more powerful than language alone in eliciting emotion, is processed throughout spinal, subcortical, and cortical regions, and thus has meaningful impacts on complex cognitive and affective processes. While music and language utilize similar features in the brain, music is more rooted in the primitive brain structures involved in motivation, reward, and emotion. Within the brain, emotional, language, and memory centers are connected during music processing.

Theoretical/Conceptual Framework

Two complementary models guide this study: The Dual-Process Model of Coping with Bereavement and the Meaning Reconstruction Model. Both models view grief as a life-long process of renegotiating continuing bonds with the deceased and finding meaning in life after the loss. The dual-process model posits that grieving a loved one entails oscillating between orientation to the loss (i.e., continuing bonds with the deceased by expressing emotion related to the death and reconnecting with the memory of the loved one) and restoration of contact with a changed world (i.e., re-engaging relationships and experimenting with new life roles). The meaning reconstruction model of grief views grieving as a process of reaffirming or reforming a world of meaning that has been challenged by loss. Research on these models demonstrates signs of efficacy, particularly regarding how continuing bonds with the deceased and meaning-making are important mechanisms of successful adaption to bereavement.

Preliminary Work

This team has implemented two pilot studies examining the in-person and online delivery of STM to professional caregivers. In both studies, the intervention delivery method was feasible and significant improvements were seen in coping (self-compassion (F(3, 105) = 2.88, p<.05), self-awareness (F(3, 120) = 2.42, p<.10), psychosocial (loneliness (F(3, 98) = 7.46, p<.001), and functional (insomnia (F(3, 120) = 5.77, p<.001) well-being. Qualitatively, participants reported feeling less emotional loneliness, and the stories and songs provided reflection and meaning-making. An unexpected finding from this study was that 60% of participants in the intervention arm had experienced a significant family loss (mostly to cancer) that inspired their oncology nursing careers. During the intervention, this primary family loss, with the grief they needed to examine. This finding informed our team of the need for bereavement interventions for family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* able to read and speak English
* bereaved parent of a child who died from cancer (ages<39 years)
* child's death >6 months and <5 years before study initiation
* access to the internet and computer.

Exclusion Criteria:

* do not have the technological requirements for Zoom interviews and REDCap surveys.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Study Feasibility | Immediately post-intervention (6 weeks)
  Feasibility will be evaluated by tracking the percentage of participants screened and enrolled. The study will be deemed feasible with a 60% enrollment rate.
Intervention Feasibility | Immediately post-intervention (6 weeks)
  Feasibility will be evaluated by tracking the average number of sessions the participants complete. This intervention will be deemed feasible if 85% of the intervention is completed.
Intervention Acceptability | Immediately post-intervention (6 weeks)
  An additional primary endpoint is acceptability. Acceptability will be evaluated with semi-structured interview questions to understand the participant's perception of intervention delivery and content, as well as the perceived impact.

SECONDARY OUTCOMES:
Mean Change from Baseline in Anxiety Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short-Form 8a will be used. The minimum score is 8, and the maximum score is 40. Higher scores indicate more anxiety.
Mean Change from Baseline in Depression Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form 8a will be used.The minimum score is 8, and the maximum score is 40. Higher scores indicate higher levels of depressive symptoms.
Mean Change from Baseline in Quality of Life Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life scale (10 items) will be used. The minimum score is 5, and the maximum score is 50. Higher scores indicate more sleep disturbance.
Mean Change from Baseline in Sleep Disturbance Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short-Form 6a will be used. The minimum score is 6, and the maximum score is 30. Higher scores indicate more sleep disturbance.
Mean Change from Baseline in Loneliness Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  UCLA Loneliness Scale; range is 0-60; lower score is better outcome.
Mean Change from Baseline in Self-Compassion Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  Self-Compassion Scale; range is 26-130; higher score is better outcome.
Mean Change from Baseline in Metacognition Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Metacognition Questionnaire-30; range from 30 - 120; higher score is better outcome.
Mean Change from Baseline in Continuing Bonds Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Continuing Bonds Scale; ranges from 11-55.
Mean Change from Baseline in Prolonged Grief Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Prolonged Grief-13-Revised; range 10-50; higher score means greater prolonged grief.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Phillips, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No